CLINICAL TRIAL: NCT02245737
Title: A 24-month, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Efficacy, Safety, Tolerability, Biomarker, and Pharmacokinetic Study of AZD3293 in Early Alzheimer's Disease (The AMARANTH Study)
Brief Title: An Efficacy and Safety Study of Lanabecestat (LY3314814) in Early Alzheimer's Disease
Acronym: AMARANTH
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: An independent assessment concluded the trial was not likely to meet the primary endpoint upon completion and therefore, trial stopped for futility
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16023; I8D-MC-AZES (Other: Eli Lilly and Company); 2014-002601-38 (EudraCT Number); D5010C00009 (Other: AstraZeneca)
Record Dates: First submitted 2014-09-18; First posted 2014-09-22 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer´s Disease
Keywords: Alzheimer's disease; Dementia; Brain Diseases; Neurogenerative Diseases; Central Nervous System Diseases; Nervous System Diseases; Mental Disorders; Delirium, Dementia, Amnestic, Cognitive Disorders; Tauopathies
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Mental Disorders; Neurocognitive Disorders; Tauopathies | interventions — lanabecestat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lanabecestat 20 milligrams (mg) (Experimental): Lanabecestat 20 mg given orally once daily for 104 weeks.
  Interventions: Drug: Lanabecestat
- Lanabecestat 50 mg (Experimental): Lanabecestat 50 mg given orally once daily for 104 weeks.
  Interventions: Drug: Lanabecestat
- Placebo (Placebo Comparator): Placebo given orally once daily for 104 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lanabecestat — Administered orally
  Other Names: LY3314814; AZD3293
  Arms: Lanabecestat 20 milligrams (mg); Lanabecestat 50 mg
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of lanabecestat compared with placebo administered for 104 weeks in the treatment of early Alzheimer´s disease. The study will test the hypothesis that lanabecestat is a disease-modifying treatment for participants with early Alzheimer´s disease, defined as the continuum of participants with mild cognitive impairment (MCI) due to Alzheimer´s disease and participants diagnosed with mild dementia of the Alzheimer´s type, as measured by change from baseline on the 13-item Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13) score at week 104 in each of the 2 lanabecestat treatment groups compared with placebo.

DETAILED DESCRIPTION:
Participants who meet other study entry requirements will be required to undergo either an amyloid positron emission tomography (PET) scan or a lumbar puncture for cerebrospinal fluid (CSF) sampling at screening to document presence of abnormal levels of brain and CSF amyloid for study inclusion. The study includes 2 sub-studies: the participants that undergo a PET scan at screening will be included in the PET-substudy, and participants who undergo a lumbar puncture at screening will be included in the CSF substudy until each of these substudies are completed.

ELIGIBILITY:
Inclusion Criteria:

* Gradual and progressive change in the participant's memory function over more than 6 months, reported by participant and study partner
* Mini-Mental State Examination score of 20-30 inclusive at screening
* Objective impairment in memory as evaluated by memory test performed at screening
* For a diagnosis of mild Alzheimer's Disease (AD), participant meets the National Institute on Aging and the Alzheimer's Association (NIA-AA) criteria for probable AD
* For a diagnosis of MCI due to AD, participant meets NIA-AA criteria for MCI due to AD

Exclusion Criteria:

* Significant neurological disease affecting the central nervous system, other than AD, that may affect cognition or ability to complete the study, including but not limited to, other dementias, serious infection of the brain, Parkinson´s disease, or epilepsy or recurrent seizures
* History of clinically evident stroke, or multiple strokes based on history or imaging results
* History of clinically important carotid or vertebrobasilar stenosis or plaque
* History of multiple concussions with sustained cognitive complaints or objective change in neuropsychological function in the last 5 years
* Participants with a current Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition diagnosis of Major Depressive Disorder or any current primary psychiatric diagnosis other than AD if, in the judgment of the investigator, the psychiatric disorder or symptom is likely to confound interpretation of drug effect, affect cognitive assessments, or affect the participant´s ability to complete the study
* History of alcohol or drug abuse or dependence (except nicotine dependence) within 2 years before the screening
* Within 1 year before the screening or between screening and baseline, any of the following: myocardial infarction; moderate or severe congestive heart failure, New York Heart Association class III or IV; hospitalization for, or symptom of, unstable angina; syncope due to orthostatic hypotension or unexplained syncope; known significant structural heart disease (eg, significant valvular disease, hypertrophic cardiomyopathy), or hospitalization for arrhythmia
* Congenital QT prolongation
* History of cancer within the last 5 years, with the exception of non-metastatic basal and/or squamous cell carcinoma of the skin, in situ cervical cancer, non-progressive prostate cancer or other cancers with low-risk of recurrence or spread
* Current serious or unstable clinically important systemic illness that, in the judgment of the investigator, is likely to affect cognitive assessment, deteriorate, or affect the participant's safety or ability to complete the study, including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, or hematologic disorders

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2218 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon- Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (253):
- United States (77):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - St Josephs Hospital and Medical Center, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Territory Neurology & Research Institute, Tucson, Arizona
  - Positron Research International, Fremont, California
  - Alliance Research Centers, Laguna Hills, California
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Collaborative Neuroscience Network - CNS, Long Beach, California
  - Pacific Research Network Inc, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Mile High Research Center, Denver, Colorado
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Brain Matters Research, Delray Beach, Florida
  - Direct Helpers Medical Center, Hialeah, Florida
  - Berma Research, Hialeah, Florida
  - Galiz Research, Hialeah, Florida
  - MaxBlue Institute, Hialeah, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Medical Research Center, Miami, Florida
  - Allied Biomedical Research Institute, Inc., Miami, Florida
  - Advance Medical Research Institute, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - JDH Medical Group, LLC, Miami, Florida
  - Compass Research, Orlando, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Roskamp Institute, Sarasota, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Compass Research, The Villages, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - The Multiple Sclerosis Center of Atlanta, Atlanta, Georgia
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - ActivMed Practices & Research, Inc, Methuen, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Springfield Neurology Associates, Springfield, Massachusetts
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Millennium Psychiatric Associates, LLV, St Louis, Missouri
  - St. Louis Clinical Trials, LC, St Louis, Missouri
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - AdvanceMed Research, Lawrenceville, New Jersey
  - Alzheimer's Research Company, Paterson, New Jersey
  - The Cognitive and Research Center of NJ, Springfield, New Jersey
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Neurology Specialists of Monmouth County, West Long Branch, New Jersey
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - SPRI Clinical Trials, LLC., Brooklyn, New York
  - Alzheimer's Disease and Memory Disorders Center, Buffalo, New York
  - Empire Neurology, PC, Latham, New York
  - Clinilabs, Inc (New York), New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Alzheimer's Memory Center, Charlotte, North Carolina
  - Valley Medical Primary Care, Centerville, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - The Corvallis Clinic P.C., Corvallis, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Radiant Research, Greer, South Carolina
  - Quillen College of Medicine, East TN State University, Johnson City, Tennessee
  - Senior Adults Specialty Research Inc, Austin, Texas
  - Texas Health Physicians Group, Dallas, Texas
  - Medical Group of Texas, Fort Worth, Texas
  - University of Texas Health Services Center - Houston, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - The Memory Clinic, Bennington, Vermont
- Australia (9):
  - Southern Neurology, Kogarah, New South Wales
  - Griffith University, Gold Coast, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Delmont Private Hospital, Glen Iris, Victoria
  - Heidelberg Repatriation Hospital, Heidelberg, Victoria
  - The Florey Institute of Neuroscience and Mental Health, Parkville, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
  - Neuro Trials Victoria Pty Ltd, Noble Park
- Belgium (7):
  - Jessa Ziekenhuis, Hasselt, Limburg
  - Hopital Universitaire Brugmann Brussel, Brussels
  - Hospital Universitaire Erasme Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - Heilig Hartziekenhuis, Roeselare
- Canada (15):
  - The Medical Arts Health Research Group, Kamloops, British Columbia
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - True North Clinical Research Halifax, LLC, Halifax, Nova Scotia
  - Bruyere Continuing Care, Ottawa, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - CSSS-Institut Universitaire Gériatric de Sherbrooke, Sherbrooke, Qubec
  - Clinique de la Memoire de l'Outaouais, Gatineau, Quebec
  - NeuroSearch Developements, Greenfield Park, Quebec
  - Hopital Maisonneure-Rosemount, Montreal, Quebec
  - Hopital de L'Enfant Jesus, Québec, Quebec
  - Q&T Research Sherbrooke Inc, Sherbrooke, Quebec
- France (11):
  - CHU de Toulouse Hopital Purpan, Toulouse, Cedex 9
  - Hopital Neuro Pierre Wertheimer, Bron
  - CHU Dijonon, Dijon
  - CHRU Lille - Hopital Roger Salengro, Lille
  - CHU Hopital de la Timone, Marseille
  - Chu de Nantes Hopital Laennec, Nantes
  - Hopital Broca, Paris
  - Hopital de la Pitie Salpetriere, Paris
  - Hopital Lariboisière, Paris
  - CHU de Toulouse, Toulouse
  - Hopital des Charpennes, Villeurbanne
- Germany (21):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Studien und Gedächtniszentrum München, München, Bavaria
  - Klinikum Rechts der Isar der TU München, München, Bavaria
  - Institut fur Psychogerontologie, Nuremberg, Bavaria
  - Neurozentrum Prien, Prien am Chiemsee, Bavaria
  - Institut für Neuropsychiatrie INP3, Wenzenbach, Bavaria
  - Studienzentrum Nord-West, Westerstede, Lower Saxony
  - Praxis Dr. Lauter, Bochum, North Rhine-Westphalia
  - St Josef-Hospital Bochum, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Gemeinschaftspraxis für Neurologie Prof. Gereon Nelles, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Neurologische Praxis Siegen, Siegen, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Pharmakologisches Studienzentrum Chemnitz, Mittweida, Saxony
  - Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt
  - Universitätsklinikum Otto-von-Guericke-Universität, Magdeburg, Saxony-Anhalt
  - Arztpraxis Dr. Christian Oehlwein, Gera, Thuringia
  - Gemeinschaftspraxis Dr. R. Ehret & Dr. W. von Pannwitz, Berlin
  - Charité Universitätsmedizin Berlin, Berlin
- Hungary (6):
  - PTE KK Pszichiatriai es Pszichoterapias Klinika, Pécs, Baranya
  - Semmelweis Medical University, Budapest
  - Del-pesti Centrumkorház - Orszagos Hematologiai és Infektologiai Intezet, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Univerisity of Szeged, Szeged
- Italy (15):
  - Ospedale Degli Infermi ASR USSL 12, Ponderano, Biella
  - Azienda Ospedaliera San Gerardo, Monza, Milano
  - Fondazione San Raffaele Giglio di Cefalu, Cefalù, Palermo
  - Universita Di Pisa, Pisa, PI
  - Università Politecnica delle Marche Torrette, Ancona
  - IRCCS San Giovanni di Dio Fatebenefratelli, Brescia
  - Fondazione Universitaria degli Studi G D'Annunzio, Chieti
  - Ente Ospedaliero Ospedali Galliera, Genova
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policinico, Milan
  - Nuovo Ospedale Civile Sant'Agostino Estense, Modena
  - Policlinico Univ. Agostino Gemelli, Roma
  - Dip.to Med. Sperimentale -Polic.Umberto I -Univ. La Sapienza, Roma
  - Ospedale San Giovanni Calibita Fatebenefratelli, Roma
  - Policlinico Ospedale S. Andrea, Roma
  - Azienda Ospedaliera Citta della Salute della Scienza Torino, Torino
- Japan (31):
  - National Institute for Longevity Sciences NCGG, Ōbu, Aichi-ken
  - National Chiba-East-Hospital, Chuo-ku, Chiba
  - National Hospital Organization Asahikawa Medical Center, Asahikawa, Hokkaido
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Iwate Medical University Hospital, Morioka, Iwate
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Nihon Kokan Hospital, Kawasaki, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Rakuwakai Otowarehabilitation Hospital, Kyoto, Kyoto
  - Ina Central Hospital, Ina, Nagano
  - Matsumoto Medical Center, Matsumoto, Nagano
  - Katayama Medical Clinic, Kurashiki, Okayama-ken
  - Shiroma Clinic, Urasoe, Okinawa
  - Koshokai aino hospital, Ibaraki, Osaka
  - Sakaguchi Clinic, Sakai, Osaka
  - National Sanatorium Toneyama Hospital, Toyonaka, Osaka
  - Saitama Medical University Hospital, Iruma-Gun, Saitama
  - Nippon Medical School Hospital, Bunkyo-Ku, Tokyo
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - Nozomi Memory Clinic, Mitaka-shi, Tokyo
  - Sangenjaya Nakamura Mental Clinic, Setagaya City, Tokyo
  - Kanauchi Medical Clinic, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Memory Clinic Ochanomizu, Tsukuba, Tokyo
  - National Sanatorium Hokuriku Hospital, Nanto, Toyama
  - Fukuoka University Hospital, Fukuoka
  - Kyoto University Hospital, Kyoto
  - Kyoto Minami Hospital, Kyoto
  - Utano Hospital, Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
- Poland (13):
  - NZOZ Wroclawskie Centrum Alzheimerowskie, Wroclaw, Lower Silesian Voivodeship
  - Medycyna Milorzab, Lodz, Lódzkie
  - Podlaskie Centrum Psychogeriatrii, Bialystok, Podlaskie Voivodeship
  - NZOZ Dom Sue Ryder - Pallmed Sp. z o.o., Bydgoszcz
  - NZOZ Wielospecjalistyczna Poradnia Lekarska, Katowice
  - Specjalistyczna Praktyka Lekarska prof. Grzegorz Opala, Katowice
  - Centrum Zdrowia Psychicznego, Kielce
  - Centrum Neurologii Klinicznej, Krakow
  - NZOZ Neuromed M. I M. Nastaj sp. P., Lublin
  - Instytut Medycyny Wsi, Lublin
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Siemianowice Śląskie
  - Centrum Medyczne, Warsaw
  - Centralny Szpital Kliniczny MSW, Warsaw
- Puerto Rico (4):
  - Santa Cruz Behavioral PSC, Bayamón, PR
  - Instituto de Neurologia Dra. Ivonne Fraga, San Juan, PR
  - Ivonne Z. Jimenez-Velazquez, MD, Carolina
  - Michel A. Woodbury-Farina, MD., San Juan
- Romania (4):
  - SC Med Life SA, Bucharest
  - SC Centrul Medical Sana SRL, Bucharest
  - Policlinica CCBR S.R.L., Bucharest
  - SC Med Life SA, Timișoara
- South Korea (9):
  - Dong-A University Medical Center, Seogu, Busan
  - Seoul National University Bundang Hospital, Seongnam-si, Geonggi-do
  - The Catholic University of Korea-Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggido
  - Gachon University Gil Medical Center, Namdong, Incheon
  - Inha University Hospital, Incheon
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
- Spain (19):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Virgen Del Puerto, Plasencia, Caceres
  - Hospital Universitario De Getafe, Madrid, Getafe
  - Hospital Puerta De Hierro, Majadahonda, Madrid
  - Centro de Atencion Especializada (CAE) OROITU, Getxo, Vizcaya
  - Hospital del Mar, Barcelona
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Fundacion ACE-Institut Catala de Neurociences Aplicades, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Fundacion CITA Alzheimer, Donostia / San Sebastian
  - Hospital De La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Univ Sant Joan de Reus, S.A., Reus
  - Hospital Doctor Peset, Valencia
  - Hospital Universitario La Fe de Valencia, Valencia
- United Kingdom (12):
  - Plymouth Hospitals NHS Trust, Plymouth, Devon
  - Cognitive Treatment & Research Unit, Crowborough, East Sussex
  - Southern Health NHS, Southampton, Hampshire
  - MAC UK Neuroscience Ltd, Blackpool, Lancs
  - MAC Clinical Research, Stourton, Leeds
  - MAC Clinical Research, Cannock, Staffordshire
  - West London Mental Health NHS Trust, Brentford
  - Glasgow Memory Clinic, Glasgow
  - Hammersmith Hospital, London
  - Guildford Nuffield Hospital, London
  - Re-Cognition Health Ltd, London
  - MAC Clinical Research, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Chandler JM, Lansdall CJ, Ye W, McDougall F, Belger M, Toth B, Mi X, Sink KM, Atkins AS. The Alzheimer's Disease Cooperative Study - Activities of Daily Living dependence score: revision and validation of an algorithm evaluating patient dependence across the spectrum of AD severity. J Prev Alzheimers Dis. 2025 Sep;12(8):100261. doi: 10.1016/j.tjpad.2025.100261. Epub 2025 Jul 1. PMID 40603145
- [Derived] Wessels AM, Lines C, Stern RA, Kost J, Voss T, Mozley LH, Furtek C, Mukai Y, Aisen PS, Cummings JL, Tariot PN, Vellas B, Dupre N, Randolph C, Michelson D, Andersen SW, Shering C, Sims JR, Egan MF. Cognitive outcomes in trials of two BACE inhibitors in Alzheimer's disease. Alzheimers Dement. 2020 Nov;16(11):1483-1492. doi: 10.1002/alz.12164. Epub 2020 Oct 13. PMID 33049114
- [Derived] Wessels AM, Tariot PN, Zimmer JA, Selzler KJ, Bragg SM, Andersen SW, Landry J, Krull JH, Downing AM, Willis BA, Shcherbinin S, Mullen J, Barker P, Schumi J, Shering C, Matthews BR, Stern RA, Vellas B, Cohen S, MacSweeney E, Boada M, Sims JR. Efficacy and Safety of Lanabecestat for Treatment of Early and Mild Alzheimer Disease: The AMARANTH and DAYBREAK-ALZ Randomized Clinical Trials. JAMA Neurol. 2020 Feb 1;77(2):199-209. doi: 10.1001/jamaneurol.2019.3988. PMID 31764959
- [Derived] Cebers G, Alexander RC, Haeberlein SB, Han D, Goldwater R, Ereshefsky L, Olsson T, Ye N, Rosen L, Russell M, Maltby J, Eketjall S, Kugler AR. AZD3293: Pharmacokinetic and Pharmacodynamic Effects in Healthy Subjects and Patients with Alzheimer's Disease. J Alzheimers Dis. 2017;55(3):1039-1053. doi: 10.3233/JAD-160701. PMID 27767991
- See also: Click here for more information about this study: An Efficacy and Safety Study of LY3314814 in Early Alzheimer's Disease — https://www.lillytrialguide.com/en-US/studies/mild-alzheimer-s-disease/AZES#?postal=
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=16023&attachmentIdentifier=f8802097-b8c3-4396-ad08-8df8ca98325d&fileName=CSP_NCT02245737.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=16023&attachmentIdentifier=5c8b319d-5e9f-4b1d-b366-d589b53774a8&fileName=SAP_NCT02245737.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo film-coated oral tablets once daily.
- Lanabecestat 20 Milligrams (mg): Participants received lanabecestat 20 mg film-coated oral tablets once daily.
- Lanabecestat 50 mg: Participants received lanabecestat 50 mg film-coated oral tablets once daily.
Period: Overall Study
Arm/Group | Placebo | Lanabecestat 20 Milligrams (mg) | Lanabecestat 50 mg
Started | 740 | 739 | 739
Received at Least 1 Dose of Study Drug | 738 | 736 | 735
Completed | 187 | 184 | 168
Not Completed | 553 | 555 | 571
Not completed — Adverse Event | 23 | 26 | 33
Not completed — Condition Worsened | 9 | 10 | 9
Not completed — Death | 2 | 4 | 4
Not completed — Eligibility Criteria No Longer Met | 2 | 4 | 4
Not completed — Initiation of Symptomatic AD medication | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 5 | 4
Not completed — Other-determined by Investigator | 9 | 10 | 10
Not completed — Physician Decision | 6 | 3 | 6
Not completed — Protocol Violation | 3 | 2 | 3
Not completed — Withdrawal by Subject | 40 | 41 | 44
Not completed — Withdrawal due to Caregiver Circumstance | 10 | 20 | 22
Not completed — Sponsor Decision | 445 | 430 | 432

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Lanabecestat 20 mg: Participants received lanabecestat 20 mg film-coated oral tablets once daily.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg | Total
Number analyzed (Participants) | 740 | 739 | 739 | 2218
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.4 (6.9) | 71.2 (7.5) | 71.2 (7.0) | 71.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 398 | 395 | 384 | 1177
  Male | 342 | 344 | 355 | 1041
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 26 | 24 | 93
  Not Hispanic or Latino | 626 | 650 | 644 | 1920
  Unknown or Not Reported | 71 | 63 | 71 | 205
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 85 | 85 | 102 | 272
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 6 | 16
  White | 598 | 609 | 593 | 1800
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 52 | 40 | 38 | 130
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 13 | 11 | 12 | 36
  Romania | 1 | 2 | 2 | 5
  Hungary | 7 | 12 | 6 | 25
  United States | 171 | 171 | 179 | 521
  Japan | 48 | 57 | 78 | 183
  United Kingdom | 85 | 87 | 78 | 250
  Spain | 74 | 77 | 65 | 216
  Canada | 58 | 59 | 63 | 180
  South Korea | 30 | 24 | 16 | 70
  Belgium | 20 | 15 | 15 | 50
  Poland | 58 | 51 | 50 | 159
  Italy | 45 | 38 | 49 | 132
  Australia | 38 | 55 | 38 | 131
  France | 45 | 36 | 36 | 117
  Germany | 47 | 44 | 52 | 143
ADAS-Cog13 (13-item Alzheimer's Disease Assessment Scale) [Mean (Standard Deviation); unit: Units on a Scale] — ADAS-Cog13, a 13-item rating scale, measured the severity of cognitive dysfunction in persons with Alzheimer's disease (AD). Scores ranged from 0 to 85, with a higher score indicating worse cognitive functioning.
  Units on a Scale | 28.6 (7.9) | 29.0 (7.7) | 28.5 (8.2) | 28.7 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the 13-item Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13)
Description: ADAS-Cog13 (13-item version of ADAS-Cog) is a psychometric instrument that evaluates word recall, ability to follow commands, constructional praxis, naming, ideational praxis, orientation, word recognition, memory, comprehension of spoken language, word-finding, and language ability, with a measure of delayed word recall and concentration/ distractibility. The total score of the 13-item scale ranges from 0 to 85, with an increase in score indicating cognitive worsening. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with factors for treatment, visit, treatment-by-visit interaction, disease status at baseline, apolipoprotein E4 (APOE4) status, acetylcholinesterase inhibitor (AChEI) use at baseline, pooled country, and covariates for baseline ADAS-Cog13 total score, age at baseline, and baseline ADAS-Cog13 total score-by-visit interaction.
Time Frame: Baseline, Week 104
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for ADAS-Cog13 measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 723 | 722 | 708
Units on a scale | 10.31 (0.55) | 9.38 (0.56) | 10.72 (0.58)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.232, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-2.447 to 0.594], Standard Error of Mean 0.77
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.599, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-1.124 to 1.947], Standard Error of Mean 0.78

2. Secondary Outcome: Change From Baseline on the Alzheimer´s Disease Cooperative Study Activities of Daily Living Inventory Instrumental Items (ADCS-iADL)
Description: The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-ADL measures both basic and instrumental activities of daily living by participants. The range for the ADCS-iADL is 0-59 with higher scores reflecting better performance. LS Mean was determined by MMRM model with factors for treatment, visit, treatment-by-visit interaction, disease status at baseline, APOE4 status, AChEI use at baseline, pooled country, and covariates for baseline for baseline iADL score, age at baseline, and baseline iADL score-by-visit interaction.
Time Frame: Baseline, Week 104
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for ADCS-iADL measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 702 | 700 | 674
Units on a scale | -8.87 (0.60) | -8.84 (0.61) | -8.79 (0.63)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.971, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-1.609 to 1.669], Standard Error of Mean 0.83
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.923, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-1.580 to 1.743], Standard Error of Mean 0.85

3. Secondary Outcome: Change From Baseline on the Functional Activities Questionnaire (FAQ) Score
Description: FAQ is a 10-item, caregiver-based questionnaire and was administered to the study partner who was asked to rate the participant's ability to perform a variety of activities ranging from writing checks, assembling tax records, shopping, playing games, food preparation, traveling, keeping appointments, traveling out of neighborhood, keeping track of current events and understanding media. FAQ total score was calculated by adding the scores from each of the 10 items. Each activity is rated on a scale from 0 to 3 (Never did and would have difficulty now = 1; Never did [the activity] but could do now = 0; Normal = 0; Has difficulty but does by self = 1; Requires assistance = 2; Dependent = 3). FAQ scale is 0 to 30, with higher scores indicating greater impairment. LS Mean was calculated by MMRM with factors for treatment, visit, treatment-by-visit interaction, disease status at baseline, APOE4 status, AChEI use at baseline and pooled country.
Time Frame: Baseline, Week 104
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for FAQ score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 699 | 697 | 674
Units on a scale | 6.09 (0.38) | 5.96 (0.39) | 6.71 (0.40)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.796, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-1.172 to 0.899], Standard Error of Mean 0.53
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.252, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-0.437 to 1.660], Standard Error of Mean 0.53

4. Secondary Outcome: Change From Baseline on the Integrated Alzheimer's Disease Rating Scale (iADRS) Score
Description: The iADRS is a composite that measures both cognition and function. The iADRS comprises scores form the ADAS- Cog and the ADCS-iADL. The iADRS is calculated as a linear combination of the total scores of the ADAS-Cog13 (score range 0 to 85 with higher scores reflecting worse performance) and the ADCS-iADL (score range from 0-59 with higher scores reflecting better performance). The iADRS score ranges from 0 to 144 with higher scores indicating greater impairment. LS Mean was determined by MMRM methodology with factors for treatment, visit, treatment-by- visit interaction, disease status at baseline, APOE4 status, AChEI use at baseline, pooled country, and covariates for baseline iADRS13 total score, age at baseline, and baseline iADRS13 total score-by-visit interaction.
Time Frame: Baseline, Week 104
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for iADRS.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 696 | 689 | 662
Units on a scale | -19.56 (0.99) | -18.45 (1.02) | -19.69 (1.05)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.428, Mixed Models Analysis; LS Mean Difference (Final Values) = 1.11, 95% CI 2-sided [-1.637 to 3.852], Standard Error of Mean 1.40
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.926, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-2.918 to 2.655], Standard Error of Mean 1.42

5. Secondary Outcome: Change From Baseline on the Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score
Description: The CDR-SB is a rater administered scale and impairment is scored in of the following categories: memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care. Impairment is scored on a scale in which no dementia = 0, questionable dementia = 0.5, mild dementia = 1, moderate dementia = 2 and severe dementia = 3. The 6 individual category ratings, or "box scores", were added together to give the CDR-Sum of Boxes which ranges from 0-18, with higher scores indicating greater impairment. LS Mean was determined by MMRM methodology with factors for treatment, visit, treatment-by-visit interaction, disease status at baseline, APOE4 status, AChEI use at baseline, pooled country, and covariates for baseline CDR-SB score, age at baseline, and baseline CDR-SB score-by-visit interaction.
Time Frame: Baseline, Week 104
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for CDR-SB.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 704 | 705 | 676
Units on a scale | 3.02 (0.17) | 3.17 (0.17) | 3.17 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.533, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.322 to 0.622], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.537, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.328 to 0.630], Standard Error of Mean 0.24

6. Secondary Outcome: Time to Progression as Measured by Loss of Clinical Dementia Rating (CDR) Global Score Stage
Description: The CDR global score is a composite score calculated using the Washington University CDR-assignment algorithm applied to the 6 individual domain box scores (Morris 1993). The memory domain is considered the primary category that drives the CDR global outcome, and all other domains are secondary. The CDR global score ranges from 0 to 3 (0 = no dementia, 0.5 = questionable dementia, 1 = mild dementia, 2 = moderate dementia, 3 = severe dementia).
Time Frame: Baseline through Loss of 1 Global Stage or Week 104
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for CDR Global Score.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 716 | 714 | 696
Days | 548 [547 to 554] | 547 [545 to 550] | 548 [545 to 553]

7. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Score
Description: The NPI is a questionnaire administered to caregivers that quantifies behavioral changes. Each of the 12 behavioral domains the caregiver reports as present are scored for Frequency, scale: 1 (Occasionally) to 4 (Very Frequently), and Severity, scale: 1 (Mild) to 3 (Severe). If the domain is reported by the caregiver as 'Not Affected,' that domain is scored as 0. The individual domain scores are calculated by multiplying the frequency times the severity for each domain. NPI Total Score is calculated by adding the individual domain scores together for all 12 domains, with a scores range from 0 to 144, with higher scores indicating greater severity of neuropsychiatric disturbance. LS Mean was determined by MMRM methodology with factors for treatment, visit, treatment-by-visit interaction, disease status at baseline, APOE4 status, AChEI use at baseline, pooled country, and covariates for baseline NPI score, age at baseline, and baseline NPI score-by-visit interaction.
Time Frame: Baseline, Week 104
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for NPI.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 697 | 695 | 663
Units on a scale | 3.22 (0.81) | 4.99 (0.83) | 4.67 (0.85)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.116, Mixed Models Analysis; LS Mean Difference (Final Values) = 1.77, 95% CI 2-sided [-0.441 to 3.986], Standard Error of Mean 1.13
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.208, Mixed Models Analysis; LS Mean Difference (Final Values) = 1.45, 95% CI 2-sided [-0.808 to 3.704], Standard Error of Mean 1.15

8. Secondary Outcome: Change From Baseline on the Mini-Mental State Examination (MMSE)
Description: The MMSE is an instrument used to assess a participant's global cognitive function. The MMSE assesses orientation to time and place, immediate and delayed recall of words, attention and calculation, language (naming, comprehension and repetition), and spatial ability (copying a figure). The range for MMSE total Score is 0 to 30, with a higher score indicating better cognitive performance. LS mean was determined by MMRM methodology with factors for treatment, visit, treatment-by-visit interaction, disease status at baseline, APOE4 status, AChEI use at baseline, pooled country, and covariates for baseline MMSE total score, age at baseline, and baseline MMSE total score-by-visit interaction.
Time Frame: Baseline, Week 104
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for MMSE.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 723 | 725 | 709
Units on a scale | -5.50 (0.26) | -5.18 (0.26) | -5.49 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.379, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.391 to 1.027], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.992, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.714 to 0.721], Standard Error of Mean 0.37

9. Secondary Outcome: Pharmacodynamics (PD): Percent Change From Baseline in Concentration of Cerebrospinal Fluid (CSF) Biomarker Amyloid Beta (Aβ)1-42
Description: Concentration of the peptide Aβ 1-42 in plasma measured by validated immunoassay. LS Mean was determined by Analysis of covariance (ANCOVA) with last observation carried forward (LOCF), terms for treatment, baseline biomarker and age at baseline.
Time Frame: Baseline, Week 97
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for Aβ1-42.
Measure: Least Squares Mean (Standard Error); unit: Percent change in Aβ1-42
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 63 | 66 | 79
Percent change in Aβ1-42 | -2.64 (2.07) | -53.91 (2.04) | -68.13 (1.87)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = -51.27, 95% CI 2-sided [-56.963 to -45.578], Standard Error of Mean 2.89
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = -65.48, 95% CI 2-sided [-70.947 to -60.022], Standard Error of Mean 2.77

10. Secondary Outcome: PD: Percent Change From Baseline in Concentration of CSF Biomarker Aβ1-40
Description: Concentration of the peptide Aβ 1-40 in plasma measured by immunoassay. LS Mean was determined by ANCOVA with LOCF (last observation carried forward), terms for treatment, baseline biomarker and age at baseline.
Time Frame: Baseline, Week 97
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for Aβ1-40.
Measure: Least Squares Mean (Standard Error); unit: Percent change in Aβ1-40
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 64 | 66 | 79
Percent change in Aβ1-40 | -1.92 (1.77) | -59.90 (1.74) | -75.17 (1.60)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = -57.99, 95% CI 2-sided [-62.865 to -53.108], Standard Error of Mean 2.47
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = -73.25, 95% CI 2-sided [-77.926 to -68.575], Standard Error of Mean 2.37

11. Secondary Outcome: Change From Baseline in CSF Total Tau
Description: Cerebrospinal fluid samples are collected for analysis of concentration total tau. LS Mean was determined by ANCOVA with LOCF and with factors for treatment, disease status at baseline, baseline biomarker and age at baseline.
Time Frame: Baseline, Week 97
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for CSF Total Tau.
Measure: Least Squares Mean (Standard Error); unit: Picogram per milliliter (pg/mL)
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 64 | 66 | 79
Picogram per milliliter (pg/mL) | 12.39 (8.05) | -7.48 (8.01) | -2.92 (7.30)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.081, ANCOVA; LS Mean Difference (Final Values) = -19.87, 95% CI 2-sided [-42.210 to 2.464], Standard Error of Mean 11.33
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.157, ANCOVA; LS Mean Difference (Final Values) = -15.31, 95% CI 2-sided [-36.555 to 5.938], Standard Error of Mean 10.78

12. Secondary Outcome: Change From Baseline in CSF Phosphorylated Tau
Description: Cerebrospinal fluid samples are collected for analysis of concentrations of phosphorylated tau. LS Mean was determined by ANCOVA with LOCF and with factors for treatment, disease status at baseline, baseline biomarker and age at baseline.
Time Frame: Baseline, Week 97
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for CSF Phosphorylated Tau.
Measure: Least Squares Mean (Standard Error); unit: Picogram per milliliter (pg/mL)
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 63 | 66 | 79
Picogram per milliliter (pg/mL) | 0.47 (0.95) | -2.16 (0.94) | -1.66 (0.85)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.050, ANCOVA; LS Mean Difference (Final Values) = -2.62, 95% CI 2-sided [-5.243 to -0.002], Standard Error of Mean 1.33
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.095, ANCOVA; LS Mean Difference (Final Values) = -2.12, 95% CI 2-sided [-4.618 to 0.373], Standard Error of Mean 1.27

13. Secondary Outcome: Change From Baseline in Brain Amyloid Burden Using Florbetapir Amyloid Positron Emission Tomography (PET) Scan
Description: Amyloid deposition in the brain is one of the defining neuropathologic findings of Alzheimer's disease. Florbetapir exhibits high affinity specific binding to amyloid plaques. The change from baseline was measured as average standard uptake value ratio (SUVr) in prespecified regions of interest (ROI) assessed by florbetapir amyloid PET imaging in a subset of participants. The Centiloid scale standardizes quantitative brain amyloid PET results to allow cross-tracer and cross-methodology comparisons. The Centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scans. Florbetapir SUVr was converted to the Centiloid scale using the following conversion: Florbetapir Centiloids = 183 x SUVr - 177. LS Mean was determined by ANCOVA methodology with factors for treatment, disease status at baseline, baseline biomarker and age at baseline.
Time Frame: Baseline, Week 104
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for brain amyloid burden.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 133 | 127 | 116
Units on a scale | -2.08 (1.86) | -15.76 (1.89) | -19.74 (1.97)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = -13.68, 95% CI 2-sided [-18.785 to -8.574], Standard Error of Mean 2.60
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = -17.66, 95% CI 2-sided [-22.887 to -12.428], Standard Error of Mean 2.66

14. Secondary Outcome: Change From Baseline in Tau PET ((Flortaucipir F18)
Description: Tau PET tracer (flortaucipir F18) longitudinal study measured whether lanabecestat, in participants with mild AD dementia, affected tau density and distribution over time. The outcome reported is the composite summary of the standard uptake value ratio (SUVR) normalized to the signal intensity in white matter. Annualized change is derived as change at LOCF divided by (LOCF date - baseline date) multiplied by 365. LS Mean was determined by ANCOVA methodology with factors for treatment, disease status at baseline, baseline biomarker and age at baseline. Baseline defined to be within 28 days of starting study drug.
Time Frame: Baseline, Week 104
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for Tau PET.
Measure: Least Squares Mean (Standard Error); unit: Standard Uptake Value ratio (SUVr)
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 97 | 94 | 93
Standard Uptake Value ratio (SUVr) | 0.04 (0.01) | 0.03 (0.01) | 0.03 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.426, ANCOVA; LS Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.033 to 0.014], Standard Error of Mean 0.01
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.660, ANCOVA; LS Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.029 to 0.018], Standard Error of Mean 0.01

15. Secondary Outcome: Change From Baseline in Brain Metabolism Using Fluorodeoxyglucose (FDG)
Description: Fluorodeoxyglucose (FDG) PET evaluates the regional brain metabolic rates for glucose as a sensitive, in vivo metabolic index of brain function. The outcome reported is the composite summary of the standard uptake value ratio (SUVR) normalized to the pons + vermis assessed with composite meta and composite meta automated anatomical labeling atlas (ALL). Annualized change is derived as change at LOCF divided by (LOCF date - baseline date) multiplied by 365. LS Mean was determined by ANCOVA methodology with factors for treatment, disease status at baseline, baseline biomarker and age at baseline. Baseline defined to be within 28 days of starting study drug.
Time Frame: Baseline, Week 104
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data of brain metabolism.
Measure: Least Squares Mean (Standard Error); unit: Standard Uptake Value ratio (SUVr)
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 83 | 95 | 82
Standard Uptake Value ratio (SUVr) | -0.04 (0.00) | -0.05 (0.00) | -0.05 (0.00)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.210, ANCOVA; LS Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.015 to 0.003], Standard Error of Mean 0.00
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.568, ANCOVA; LS Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.013 to 0.007], Standard Error of Mean 0.00

16. Secondary Outcome: Change From Baseline in Whole Brain Volume
Description: Magnetic resonance imaging (MRI) was used to evaluate the effect of lanabecestat on whole brain volumes. Annualized change is derived as change at LOCF divided by (LOCF date - baseline date) multiplied by 365. LS Mean was determined by ANCOVA methodology with factors for treatment, baseline vMRI, intracranial volume, disease status at baseline and age at baseline.
Time Frame: Baseline, Week 104
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for Whole Brain Volume.
Measure: Least Squares Mean (Standard Error); unit: cm^3 (cubic centimeter)
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 565 | 582 | 550
cm^3 (cubic centimeter) | -14.16 (0.34) | -16.49 (0.33) | -17.34 (0.34)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = -2.34, 95% CI 2-sided [-3.258 to -1.413], Standard Error of Mean 0.47
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = -3.18, 95% CI 2-sided [-4.118 to -2.247], Standard Error of Mean 0.48

17. Secondary Outcome: Pharmacokinetics (PK): Plasma Concentration of Lanabecestat
Time Frame: Week 4, post dose prior to departure from the clinic
Population: All randomized participants who received at least one dose of study drug and have evaluable PK data.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 697 | 662
nanograms per milliliter (ng/mL) | 67.7 (49.1) | 213 (149)

ADVERSE EVENTS:
Time Frame: Up To 104 weeks
Description: All randomized participants who received at least one dose of study drug. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
All-Cause Mortality (participants affected / at risk) | 2/738 | 4/736 | 4/735
Serious Adverse Events (participants affected / at risk) | 108/738 | 117/736 | 147/735
Other Adverse Events (participants affected / at risk) | 340/738 | 357/736 | 361/735
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=738) | Lanabecestat 20 mg (N=736) | Lanabecestat 50 mg (N=735)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (3) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 2 (2) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Bifascicular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2) | 1 (2)
Pterygium (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Coeliac artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enlarged uvula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Femoral hernia incarcerated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 4 (4) | 4 (4)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bone abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (4)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatic cyst infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Human anaplasmosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 3 (3) | 3 (3)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Septic arthritis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (8) | 1 (1) | 3 (3)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Accidental poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Chemical burn of gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 8 (8) | 4 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 2 (2)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lacrimal structure injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 3 (4)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 5 (5)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Infrapatellar fat pad inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer male (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/341 (0) | 1/344 (1) | 0/354 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/397 (1) | 0/392 (0) | 0/381 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 3 (3)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/397 (0) | 0/392 (0) | 1/381 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/341 (2) | 2/344 (2) | 2/354 (2)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/341 (1) | 0/344 (0) | 0/354 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cholinergic syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dementia with lewy bodies (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 6 (6) | 7 (7)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Ulnar nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device failure (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Acute psychosis (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2) | 5 (5)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination, olfactory (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2/341 (2) | 1/344 (1) | 1/354 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0/397 (0) | 1/392 (1) | 0/381 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Spinal operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Synovial cyst removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Urethral repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Vocal cord operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Granulomatosis with polyangiitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=738) | Lanabecestat 20 mg (N=736) | Lanabecestat 50 mg (N=735)
Diarrhoea (Gastrointestinal disorders) | 39 (44) | 62 (81) | 54 (62)
Nausea (Gastrointestinal disorders) | 32 (38) | 33 (39) | 41 (50)
Nasopharyngitis (Infections and infestations) | 60 (69) | 78 (94) | 76 (89)
Upper respiratory tract infection (Infections and infestations) | 46 (57) | 39 (43) | 44 (50)
Urinary tract infection (Infections and infestations) | 56 (70) | 36 (53) | 32 (36)
Fall (Injury, poisoning and procedural complications) | 69 (86) | 71 (95) | 73 (111)
Back pain (Musculoskeletal and connective tissue disorders) | 40 (50) | 36 (38) | 33 (35)
Dizziness (Nervous system disorders) | 42 (48) | 43 (52) | 51 (61)
Headache (Nervous system disorders) | 52 (56) | 40 (50) | 46 (72)
Anxiety (Psychiatric disorders) | 34 (40) | 57 (63) | 48 (50)
Depression (Psychiatric disorders) | 31 (32) | 36 (39) | 46 (49)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (25) | 46 (49) | 25 (29)

LIMITATIONS AND CAVEATS:
An independent assessment concluded the trial was not likely to meet the primary endpoint upon completion and therefore, trial stopped for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor shall review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60days but less than or equal to 180days from the time submitted to the sponsor.Authors agree not to publish results until data is compiled. No publication/presentation with respect to the research activities shall be made unless & until any information determined at sponsors sole discretion to be confidential information has been removed.

DOCUMENTS (2):
  • Study Protocol (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02245737/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02245737/SAP_001.pdf